CLINICAL TRIAL: NCT00853931
Title: An Exploratory Trial of Biomarkers for Panitumumab Response Among Previously Treated Patients With KRAS Wild Type Metastatic Colorectal Cancer.
Brief Title: Biomarker - Panitumumab Response With KRAS Wild Type MCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CA-2008-0012; KRAS wild type; metastatic colorectal cancer
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: KRAS wild type; metastatic colorectal cancer; KRAS wild type metastatic colorectal cancer with no prior exposure to EGFR inhibitors
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab (Experimental): Panitumumab 6 mg/kg will be administered by intravenous infusion every 2 weeks (Q2W), +/- 3 days, (eg, week 1, 3, 5 [i.e. Cycles 1, 2, 3, etc.]) until disease progression or intolerance panitumumab as determined by the investigator.
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab — Panitumumab 6 mg/kg will be administered by intravenous infusion every 2 weeks (Q2W), +/- 3 days, (eg, week 1, 3, 5 [i.e. Cycles 1, 2, 3, etc.]) until disease progression or intolerance panitumumab as determined by the investigator.

SUMMARY:
This is an exploratory study in which all eligible subjects are given Panitumumab according to the dose and schedule approved by Health Canada. The purpose of this research study is to determine whether the presence of certain biomarkers (substances measurable in blood, normal cells or tumour tissue) are associated with an increased or decreased chance of benefit from panitumumab.

DETAILED DESCRIPTION:
Colon cancer affects 20,000 Canadians a year. Despite efforts to improve screening, 8,500 patients will die of the disease (1). The agents used in both the adjuvant and metastatic setting have dramatically changed over the past ten years. Even with the optimal treatment and careful follow-up many patients will develop metastasis. For most this is an incurable condition and the median survival for these patients is only 2 years (2).

Therapy with 5-Fluorouracil (FU)/Leucovorin, oxaliplatin and irinotecan with or without bevacizumab are conventionally used as first and second line therapy for metastatic colorectal cancer. Third line therapy options are limited to anti-epidermal growth factor receptor (EGFR) therapy Cetuximab or Panitumumab either as monotherapy or in combination with Irinotecan. Recent data (see Table 1) has demonstrated that KRAS mutation status is a predictor of benefit to anti-EGFR therapy, with wild-type tumours demonstrating a response rate of 10-17% to monotherapy while a 0% response rate is observed among KRAS mutant tumours.

The purpose of this exploratory study is to examine the correlation of biomarkers (PTEN, BRAF, amphiregulin, c-MET, EGFR) with response rate among patients with KRAS wild type tumours treated with panitumumab. If a high response subgroup can be identified, this may support the use of Panitumumab with combination therapy in the first line setting. Secondary objectives are to determine the prognostic and predictive value of CTCs for patients treated with single agent panitumumab and to describe overall survival (OS) and progression free survival (PFS) in registered patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histological proof of adenocarcinoma of colon or rectum. In addition, proof either radiologically, or histologically that there is metastatic disease.
2. Archival, paraffin embedded tumour tissue block suitable for KRAS and biomarker, or, willingness to undergo biopsy to obtain such.
3. Received a prior thymidylate synthase inhibitor (e.g. 5-fluorouracil (5- FU), capecitabine, raltitrexed) for adjuvant and/or metastatic disease. Thymidylate synthase inhibitor may have been given in combination with oxaliplatin or irinotecan.
4. Received or ineligible for irinotecan based therapy (i.e. single-agent or in combination) for metastatic disease
5. Received or ineligible for oxaliplatin based therapy for metastatic and/or adjuvant disease.
6. Measurable or evaluable disease by RECIST criteria.
7. Adequately recovered from recent surgery, chemotherapy and/or radiation therapy. At least 4 weeks must have elapsed from major surgery, prior chemotherapy, and prior treatment with an investigational agent or prior radiation therapy.
8. Must not have received any prior anti-EGFR therapies including tyrosine kinase inhibitors or monoclonal antibodies.
9. An ECOG performance status of 0, 1 or 2.
10. Hematology done within 14 days and with initial values within the ranges specified below:

    * Absolute granulocyte count (AGC) > 1.5 x 109/L
    * Platelets > 100 x 109/L
    * Hemoglobin > 100 g/L
11. Biochemistry done within 14 days and with initial values within the ranges specified below:

    * Total bilirubin < 2.5 x institutional upper limit of normal
    * ALT < 5.0 x institutional upper limit of normal
    * AST < 5.0 x institutional upper limit of normal
    * Serum creatinine < 1.5 x institutional upper limit of normal
12. Imaging investigations including chest x-ray and CT/MRI of abdomen/pelvis or other scans as necessary to document all sites of disease done within 28 days prior to randomization. Where chest x-ray is suspicious for or reveals metastatic disease, a CT/MRI scan of the chest must also be performed. A CT/MRI scan of the chest within 28 days prior to randomization may be substituted for chest x-ray.
13. ECG done within 28 days prior to enrollment
14. Patient's age is >18 years.
15. Women of child bearing potential (WOCBP) and male partners of WOCBP must agree to use adequate contraception prior to study entry, throughout the study and for a period of 6 months after cessation of protocol therapy.
16. Adequate contraception is defined as follows:

    * Complete abstinence from intercourse from four weeks prior to administration of the first dose until 6 months after the final dose of panitumumab
    * Consistent and correct use of one of the following methods of birth control: i. male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject; or ii. implants of levonorgesterol; or iii. injectable progestagen; or iv. any intrauterine device (IUD) with a documented failure rate of less than 1% per year; or v. oral contraceptive pill (either combined or progesterone only); or vi. barrier methods including diaphragm or condom with a spermicide.
17. The baseline assessment must be completed within 14 days prior to randomization.
18. Patients must be accessible for treatment and follow-up.

Exclusion Criteria:

1. Known hypersensitivity to panitumumab or any other component of the product; life-threatening infusion reactions associated with previous administration of monoclonal antibody therapy.
2. Women who are pregnant or breastfeeding, or intend to become pregnant within the study period
3. Any active pathological condition which would render the protocol treatment dangerous or impair the ability of the patient to receive protocol therapy.
4. Any condition (e.g. psychological, geographical, etc.) that does not permit compliance with the protocol.
5. Significant history of uncontrolled angina, arrhythmias, cardiomyopathy, congestive heart failure, or documented myocardial infarction within the 6 months preceding registration (pre-treatment ECG evidence only of infarction will not exclude patient).
6. Symptomatic metastases in the central nervous system.
7. A history of prior cetuximab or other therapy which targets the Epidermal Growth Factor Receptor pathway (e.g. TarcevaTM (OSI-774), IressaTM (ZD1839), or others). A history of prior murine monoclonal antibody therapy (e.g. EdrecolomabTM (MoAB17-1A), or others).
8. Severe restrictive lung disease or radiological pulmonary findings of "interstitial lung disease" on the baseline chest x-ray which, in the opinion of the investigator, represents significant pathology.
9. Receipt of an experimental therapeutic agent within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Response rate | 1 year

SECONDARY OUTCOMES:
Clinical Benefit Rate | 1 year
Progression free survival (PFS) | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hagen Kennecke, MD, Study Chair — British Columbia Cancer Agency
Locations (3):
- Canada (3):
  - BC Cancer Agency - Abbotsford, Abbotsford, British Columbia
  - BCCA- Fraser Valley, Surrey, British Columbia
  - BC Cancer Agency, Vancouver, British Columbia